CLINICAL TRIAL: NCT01460823
Title: Percutaneous Cochlear Implantation: Implementation of Technique
Acronym: PCI-I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Currently in the process of submitting IDE to the FDA
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Robert F. Labadie, Associate Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111114
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Hearing Loss
Keywords: Hearing loss; Cochlear Implantation; Image guided surgery
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Use of image guided surgery (Experimental)
  Interventions: Procedure: Percutaneous Cochlear Implantation using image guided surgical techniques

INTERVENTIONS:
Procedure: Percutaneous Cochlear Implantation using image guided surgical techniques — Percutaneous Cochlear Implantation using image guided surgical techniques.

SUMMARY:
The investigators are studying a new way of doing cochlear implant surgery called "Percutaneous Cochlear Implantation". In this surgery, instead of doing a mastoidectomy where about 30ml of bone is removed, the investigators use image-guided technology (similar to GPS systems used to guide automobile travel) to drill directly from the surface of the skull to the cochlea, removing less than 2ml of bone. To use this technique, three markers (or anchor screws) are screwed into the bone around the ear. Next, an x-ray of the head (called a CT scan) is taken. Using this CT scan, a path to the inner ear (cochlea) is planned and a drill guide (Microtable) is made that mounts on the anchor screws. A drill will be attached to the guide and used to drill a path from the surface of the skull to the inner ear (cochlea). The implant electrode will be threaded through this path. All of these procedures take place under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year old patients undergoing cochlear implantation who are able to participate in the informed consent process.
* Pre-operative CT scan of head performed as standard of care for cochlear implant work-up.

Exclusion Criteria:

* Patients with co-morbidities so severe that the potential additional operating room time is deemed to be too significant of an operative risk. This assessment is made by the local institutions pre-operative work-up.
* History of allergic reaction/intolerance of local anesthesia and/or epinephrine.
* History of allergic reaction to titanium.
* Patients with severe anatomical abnormality of the temporal bone.
* Patients with severe chronic ear disease for whom traditional mastoidectomy might offer benefit.
* Females who are pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who underwent successful Cochlear Implantation Via Percutaneous Method | Participants will be followed post operatively until their 1st follow up visit with surgeon which on average is 3 weeks after surgery.
  A successful percutaneous cochlear implantation is one where the facial nerve was not damaged during the procedure and the surgeon did not resort back to the standard implantation method. We will measure the percentage of participants who underwent successful cochlear implantation via the percutaneous method.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Labadie, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Click here for more information related to Dr. Labadie and Otology Research at Vanderbilt University Medical Center — http://www.vanderbilt.edu/CAOS/